CLINICAL TRIAL: NCT01409499
Title: A Prospective Multicenter Non-randomized Controlled Study of Palliative Treatments for Patients With Advanced Hepatocellular Carcinoma
Brief Title: Palliative Treatments for Patients With Advanced Hepatocellular Carcinoma (HCC)
Acronym: 2011PTAHCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, XU li, Department of Hepatobiliary Surgery, Cancer Center, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011PTAHCC
Record Dates: First submitted 2011-08-01; First posted 2011-08-04 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Hepatectomy; Hepatocellular Carcinoma; Sorafenib
Keywords: hepatocellular carcinoma, treatments, survival
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A, surgery (Experimental): The patients in this group will receive palliative resection of HCC, then take sorafenib as remain therapy.
  Interventions: Procedure: hepatic resection
- B, TACE (Experimental): Patients in group B will receive transcatheter hepatic arterial chemoembolization, then take sorafenib as remain therapy.
  Interventions: Procedure: transcatheter hepatic arterial chemoembolization
- C, sorafenib (Experimental): Patients in group C will receive monotherapy of sorafenib.
  Interventions: Drug: sorafenib

INTERVENTIONS:
Procedure: hepatic resection — palliative hepatectomy followed by sorafenib
  Other Names: Group A (hepatectomy)
  Arms: A, surgery
Procedure: transcatheter hepatic arterial chemoembolization — TACE followed by sorafenib
  Other Names: Group B (TACE)
  Arms: B, TACE
Drug: sorafenib — sorafenib monotherapy, 400mg Bid, continuously
  Other Names: Group C (sorafenib)
  Arms: C, sorafenib

SUMMARY:
The standard treatment choice for advanced hepatocellular carcinoma (HCC) is sorafenib, and its efficacy is limited. More active treatments were performed in patients with advanced HCC in China, which include radical hepatectomy or TACE. The study is to investigate whether the active treatment will profit survival of patients, and to evaluate the safety.

DETAILED DESCRIPTION:
This is a prospective non-randomized controlled study. Patients with advanced hepatocellular carcinoma (BCLC C stage) who underwent palliative resection or TACE followed with Sorafenib or treated by sorafenib alone will be included. The patients will be divided to group A (palliative resection plus sorafenib), group B (palliative TACE plus sorafenib), and group C (sorafenib alone). The sample size will be about 200 cases altogether.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years of age.
* Diagnosed to have advanced HCC (BCLC C stage).
* Patients who have a life expectancy of at least 12 weeks.
* Patients whose primary tumor can be resected.

Definition of resectable in this study:

* Tumor number <=2.
* If number of tumors >= 3, then all tumors were located in the same lobe.
* Without tumor invasion of the main trunk of the portal vein, or hepatic duct, or caval vein.
* Hepatocellular carcinoma with histological diagnose or clinical diagnose according to AASLD.
* No major post-operative complication.
* Patients who have an ECOG PS of 0, or 1.
* Cirrhotic status of Child-Pugh class A only.
* The following laboratory parameters:

Platelet count > 60 x 109/L Hemoglobin > 8.5 g/dL Albumin > 3.5 g/dL Total bilirubin < 25μmol/L Alanine transaminase (ALT) and AST < 2.5 x upper limit of normal Serum creatinine <1.5 x the upper limit of normal Prothrombin time (PT)<3 seconds above control.

• Patients who give written informed consent.

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC.
* History of cardiac disease.
* Active clinically serious infections (> grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* History of organ allograft.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial.
* Pregnant or breast-feeding patients.
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.
* Excluded therapies and medications, previous and concomitant: Systemic chemotherapy and target drug other than sorafenib. Antiviral treatment is allowed.
* Radiotherapy except for which done for bone metastases palliatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | anticipate 6-12 months
  defined as the time from the first treatment to death

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | anticipate 3-6 months
  defined as the time from the first treatment to the first progression disease is confirmed by radiological methods
AEs and SAEs | anticipate 6-12 months
  according to CTC AE 3.0
cost of treatments | 3 months in average
  to compare costs of different treatments

CONTACTS AND LOCATIONS:
Overall Officials: Minshan Chen, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No